CLINICAL TRIAL: NCT05103059
Title: Prognostic Value of Serum Albumin and Total Protein in Survival of Cancer Cachectic Patients
Brief Title: Role of Serum Albumin and Total Protein in Survival of Cancer Cachectic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nehal Ali Suliman, prognostic value of serum albumin and total protein in survival of cancer cachectic patients, Assiut University
Other Study IDs: cancer cachexia
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: BMI — Patients with cancer cachexia will be enrolled in the study, and the following data will be collected: age, sex, total protein, albumin, hemoglobin (Hb), white blood cell (WBC) count, neutrophil count, lymphocyte count, red blood cell (RBC) count, platelet (PLT) count, body mass index (BMI), mid-arm circumference (MAC), thickness of triceps skinfold (TSF), handgrip strength (HGS), and calf circumference (CC)

SUMMARY:
Serum albumin can indicate the onset of cancer cachexia, provide information about a patient's nutritional status, and serve as a biomarker for the prognosis of patients with cancer cachexia. However, the relationship between serum albumin levels and mortality in patients with cancer cachexia remains unclear. We aimed to examine the association of albumin and total protein with 1-year mortality in patients with cancer cachexia

DETAILED DESCRIPTION:
Cancer cachexia is defined as a multifactorial and multi-organ syndrome characterized by the loss of skeletal muscle mass (with or without loss of adipose tissue), which cannot be fully reversed by conventional nutritional support. In recent years, cancer cachexia has increasingly been seen as a systemic phenomenon that affects various organs, such as the liver and myocardial tissue. Cachexia is closely related to anorexia, inflammation, insulin resistance, and decreased protein levels, which can lead to progressive functional impairment, treatment-related complications, poor quality of life, and cancer-related death. Its pathophysiology is characterized by a negative protein and energy balance. However, there are no clear clinical guidelines to effectively combat the progressive tissue loss associated with cachexia. Cancer cachexia occurs mostly in advanced cancers, with more than half of patients with cancer having cachexia in the later stages, and >10% of patients die with or from it.

Studies have shown that cachexia can be diagnosed when weight loss in the past 12 months is ≥5%, and the physiological variables of patients match at least threeof the following five criteria: decreased muscle strength,fatigue, anorexia, low fat-free mass index (FFMI), and abnormal blood profile. Albumin and total protein are two variables that reflect an individual's nutritional status and disease severity. Additionally, albumin can serve as an indicator of the inflammatory response and is considered a highly sensitive marker of a patient's nutritional status. Serum albumin and total protein can be used to define cancer cachexia and cancer-related malnutrition; patients with cachexia have lower total protein and albumin levels than those without cachexia.5 Serum albumin may serve as a prognostic factor for treatment outcomes and compliance in patients with advanced cancer.

Although a reduction in albumin and total protein levels are associated with the diagnosis of cancer related cachexia, no studies have shown that albumin and total protein can predict mortality in patients with cancer cachexia. Here, we describe a prospective non randomized study that will be conducted to explore the association between serum albumin and total protein levels and 1-year mortality in patients with cancer cachexia .

ELIGIBILITY:
Inclusion Criteria:

* patients who will accept to participate in our study with diagnosis of cancer cachexia

Exclusion Criteria:

* patients who not fulfill criteria of cance cachexia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: weight loss in the past 12 months is ≥5%, and the physiological variables of patients match at least threeof the following five criteria: decreased muscle strength,fatigue, anorexia, low fat-free mass index (FFMI), and abnormal blood profile
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
the association between serum albumin and total protein with one year mortality in patients with cancer cachexia | baseline
  to evaluate the association between serum albumin and total protein with one year mortality in patients with cancr cachexia

SECONDARY OUTCOMES:
the association between anthropometric measures and other laboratory findings with one year mortality in patients with cancer cachexia | baseline
  to evaluate the association between anthropometric measures and other laboratory findings with one year mortality in patients with cancer cachexia

REFERENCES:
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Background] Schmidt SF, Rohm M, Herzig S, Berriel Diaz M. Cancer Cachexia: More Than Skeletal Muscle Wasting. Trends Cancer. 2018 Dec;4(12):849-860. doi: 10.1016/j.trecan.2018.10.001. Epub 2018 Oct 24. PMID 30470306
- [Background] Evans WJ, Morley JE, Argiles J, Bales C, Baracos V, Guttridge D, Jatoi A, Kalantar-Zadeh K, Lochs H, Mantovani G, Marks D, Mitch WE, Muscaritoli M, Najand A, Ponikowski P, Rossi Fanelli F, Schambelan M, Schols A, Schuster M, Thomas D, Wolfe R, Anker SD. Cachexia: a new definition. Clin Nutr. 2008 Dec;27(6):793-9. doi: 10.1016/j.clnu.2008.06.013. Epub 2008 Aug 21. PMID 18718696
- [Background] Penet MF, Bhujwalla ZM. Cancer cachexia, recent advances, and future directions. Cancer J. 2015 Mar-Apr;21(2):117-22. doi: 10.1097/PPO.0000000000000100. PMID 25815852
- [Background] Cong M, Song C, Xu H, Song C, Wang C, Fu Z, Ba Y, Wu J, Xie C, Chen G, Chen Z, Zhou L, Li T, Deng L, Xin L, Yang L, Cui J, Shi H; Investigation on Nutrition Status and Clinical Outcome of Common Cancers (INSCOC) Group. The patient-generated subjective global assessment is a promising screening tool for cancer cachexia. BMJ Support Palliat Care. 2022 May;12(e1):e39-e46. doi: 10.1136/bmjspcare-2020-002296. Epub 2020 Aug 21. PMID 32826265
- [Background] Matsuzuka T, Kiyota N, Mizusawa J, Akimoto T, Fujii M, Hasegawa Y, Iwae S, Monden N, Matsuura K, Onozawa Y, Hayashi R, Tahara M; Japan Clinical Oncology Group(JCOG) Head and Neck Cancer Study Group. Clinical impact of cachexia in unresectable locally advanced head and neck cancer: supplementary analysis of a phase II trial (JCOG0706-S2). Jpn J Clin Oncol. 2019 Jan 1;49(1):37-41. doi: 10.1093/jjco/hyy145. PMID 30364985